CLINICAL TRIAL: NCT04277780
Title: Reducing E.D. Visits and Hospital Readmissions, and Improving Glucose Control of Patients With Uncontrolled Type 2 Diabetes by Use of Continuous Glucose Monitoring Sensors Placed at Hospital Discharge.
Brief Title: Reducing Emergency Department Visits and Improving Glucose Control in Uncontrolled Type 2 Diabetes Using CGM Sensors at Hospital Discharge
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting and following more patients during Covid-19 pandemic
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Catherine Anastasopoulou, MD, PhD, FACE, Endocrine Chair, Einstein Healthcare Network, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5100
Record Dates: First submitted 2019-04-10; First posted 2020-02-20 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: continuous glucose monitoring sensors; hospital readmission
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 70 patients assigned to intervention group (to receive CGM sensor + conventional diabetes management); 70 patients assigned to control group (to receive only conventional diabetes management)
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis to be performed on the primary and secondary outcome measure data will be provided to the assessor without information indicating whether or not a subject received the CGM sensor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM Sensor (Experimental): Subjects will receive the Libre Pro Freestyle continuous glucose monitor (CGM) sensor that will be applied to their upper arm at the time of hospital discharge. They will be asked to peel off the sensor after 14 days and mail it to the endocrinology clinic in a stamped envelope that will be provided. They will also be provided the conventional diabetes management which will include instructions on fingerstick blood glucose monitoring and logging which they will start after the CGM sensor is removed. The sensor data will be analyzed by a clinician who will call the subject regarding any changes to their diabetes management. The subject will then be asked to follow-up at the endocrinology clinic 1-month, 3-month, and 6-month from the time the sensor is placed for further management of their diabetes.
  Interventions: Device: Continuous Glucose Monitoring Sensor; Other: Diabetes Management Instructions
- Conventional Diabetes Care (Active Comparator): Subjects will receive only the conventional diabetes management at the time of hospital discharge which includes instruction on fingerstick blood glucose monitoring and logging onto a blood glucose log sheet for 14 days. They will then be asked to fax/mail/call-in the blood glucose log. The log data will be analyzed by a clinician who will call the subject regarding any changes to their diabetes management. The subject will then be asked to follow-up at the endocrinology clinic 1-month, 3-month, and 6-month from the time of hospital discharge for further management of their diabetes.
  Interventions: Other: Diabetes Management Instructions

INTERVENTIONS:
Device: Continuous Glucose Monitoring Sensor — Placement of continuous glucose monitor sensor for 14 days. Instructions on how to peel off the sensor and mail it back to the clinician.
  Arms: CGM Sensor
Other: Diabetes Management Instructions — Instructions on checking fingerstick blood glucose and information on the required equipment including glucose test strips, lancets, and glucometer. Instructions on how to log blood glucose values onto the blood glucose log sheet for 14 days, and how to mail it back to the clinician.

SUMMARY:
Quality measures and cost-reduction methods are a high priority in the United States health care system. This includes the high burden of patients with uncontrolled Type 2 Diabetes. Innovative ways to better understand and implement diabetes management plans to reduce the burden of this disease on the system are a necessity. Use of FDA-approved continuous glucose monitoring (CGM) sensors have shown benefit in better management plans in the outpatient setting. Hence, this study hypothesizes that using CGM sensors starting in the inpatient setting will provide better and quicker understanding of the disease to make expedited changes to management plans thereby improving blood glucose control and mitigating some of the health care burden by means of reducing E.D visits and hospital re-admission rates. The study will randomly assign patients to either receive a CGM sensor plus the standard diabetes management and instructions or who will only receive the standard diabetes management. The patients will be followed in the outpatient endocrinology clinic 1-month, 3-month, and 6-month from the time of hospital discharge.

DETAILED DESCRIPTION:
Rationale: Quality measures and cost-reduction methods are a high priority in the United States health care system currently. This includes the high burden of patients with uncontrolled Type 2 Diabetes on the system especially given the continued dramatic rise in the prevalence of these patients. Innovative ways to better understand and implement diabetes management plans to reduce the burden of this disease on our health care system are a necessity. The use of continuous glucose monitoring (CGM) sensors have already shown benefit in better management plans in the outpatient setting. Hence, this study aims to assess the use of CGM sensors starting in the inpatient setting and whether they will help provide better and quicker understanding of the disease to make expedited changes to management plans thereby improving blood glucose control and mitigating some of the health care burden by means of reducing E.D visits and hospital re-admission rates.

Objectives: To determine whether the use of CGM sensors in patients with uncontrolled type 2 diabetes at the time of hospital discharge leads to improved glucose control and a reduction of E.D visits and hospital readmission rates.

Trial Design: The trial design will be a randomized, non-blinded prospective study; a 1:1 comparison of uncontrolled type 2 diabetes patients who receive CGM sensors + conventional diabetes management at the time of discharge versus uncontrolled type 2 diabetes patients who receive only the conventional diabetes management.

Study Setting: Study setting will be at the Albert Einstein Medical Center (AEMC), Philadelphia, Pennsylvania for the inpatient type 2 diabetes population who will be followed at the AEMC endocrinology clinics.

ELIGIBILITY:
Inclusion Criteria:

* inpatient uncontrolled Type 2 Diabetes patients defined by HbA1c of ≥9.0% within the last 2-3 months
* require an endocrinology consultation
* will be followed at AEMC endocrinology clinic

Exclusion Criteria:

* patients with HbA1c <9.0%
* patients not managed by AEMC endocrinology clinic
* Type 1 Diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Measured at the 180-day interval post-intervention
  The difference of the average changes in HbA1c from baseline between each group (intervention vs control)
# of E.D. visits | Within 30 days from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  Number of ED visits after the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
# od hospital re-admissions | Within 30 days from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  Number of hospital re-admissions after the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data

SECONDARY OUTCOMES:
Time till first E.D. Visit | data collected for any visit occuring within 180-days from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  Length of time until first E.D. visit from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
Diabetes Mellitus (DM) Management change based on CGM sensor/log data | assessed within 30 days from the time the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  % of patients whose diabetes management was changed based on CGM sensor data or blood glucose log
Time till first hypoglycemic event | Data collected for any event occuring within 180-days from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  Time till first hypoglycemic from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
HbA1c <9.0% at the end of study | Assessed at the 180-day interval from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  # of patients with a HbA1c <9.0% at the end of the study compared to baseline
Outpatient Visit Compliance | assessed at the 180-day interval from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  % of patients who kept their outpatient clinic visits for diabetes (compliance)
Severity of first hypoglycemic event | data collected for any event occuring within 180-days from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data
  Severity of first hypoglycemic event (based on self-management vs. need call to paramedics) from the time of the first recommendation made by the clinician based on the CGM sensor data/blood glucose log data

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Anastasopoulou, MD, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No